CLINICAL TRIAL: NCT00418938
Title: A Multi-center, Open-label, Randomized, Phase 2 Clinical Trial Evaluating Safety and Efficacy of FOLFIRI With Either Panitumumab or Bevacizumab as Second-Line Treatment in Subjects With Metastatic Colorectal Cancer With Wild-type KRAS Tumors
Brief Title: SPIRITT - Second-Line Panitumumab Irinotecan Treatment Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060141
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-09

CONDITIONS: Cancer; Colon Cancer; Colorectal Cancer; Metastatic Cancer; Rectal Cancer; Metastatic Colorectal Cancer
Keywords: EGFR; FOLFIRI; 2nd Line Therapy; 2nd Line mCRC Therapy; mCRC; Irinotecan; panitumumab; bevacizumab
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis; Rectal Neoplasms | interventions — Panitumumab; Bevacizumab; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): FOLFIRI + Panitumumab
  Interventions: Drug: Panitumumab; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-Fluorouracil
- Arm B (Experimental): FOLFIRI + Bevacizumab
  Interventions: Drug: Bevacizumab; Drug: Leucovorin; Drug: Irinotecan; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Panitumumab — 6mg/kg IV
  Arms: Arm A
Drug: Bevacizumab — Either 5mg/kg OR 10mg/kg IV
  Arms: Arm B
Drug: Leucovorin — 400mg/m^2 IV (in the vein)
Drug: Irinotecan — 180mg/m^2 IV (in the vein)
Drug: 5-Fluorouracil — 400mg/m^2 bolus IV (in the vein) over 2-4 min, followed by 2400mg/m^2 continuous IV over 46 hours for the first 2 cycles, increased to 3000mg/m^2 thereafter if no significant side effects

SUMMARY:
This is a multi-center, open-label, randomized, phase 2, two-arm clinical trial to be conducted in the United States. Approximately 210 eligible KRAS wild-type expressing metastatic colorectal cancer subjects who have failed first-line oxaliplatin-based chemotherapy (with at least 4 doses of oxaliplatin-based chemotherapy) with at least 4 doses of bevacizumab (failure is defined as toxicity due to oxaliplatin-based chemotherapy or progression of disease on first-line treatment) will be randomized in a 1:1 ratio to receive either a once-every-two-weeks (Q2W) FOLFIRI regimen plus panitumumab 6 mg/kg or a Q2W FOLFIRI regimen plus bevacizumab (either 5 mg/kg or 10 mg/kg, depending on physician choice and institutional standard of care).

DETAILED DESCRIPTION:
This phase 2, multicenter, open-label, randomized, two-arm study was designed to estimate the treatment effect of panitumumab in combination with FOLFIRI compared to bevacizumab in combination with FOLFIRI in subjects with metastatic colorectal cancer (mCRC) who had failed first-line therapy with at least 4 doses of oxaliplatin-based chemotherapy and bevacizumab. After data became available demonstrating that the treatment effect of antiepidermal growth factor receptor (EGFR) agents was limited to patients with wild-type Kirsten rat Sarcoma-2 virus (KRAS) mCRC, the study was amended to enroll only subjects with wild-type KRAS tumors. Eligible subjects were randomized in a 1:1 ratio to receive panitumumab 6 mg/kg plus FOLFIRI once every 2 weeks (Q2W) or bevacizumab 5 mg/kg or 10 mg/kg plus FOLFIRI Q2W. Randomization was stratified by the reason for first-line treatment failure (progression vs toxicity) and by intended bevacizumab dose (5 mg/kg vs 10 mg/kg). The intended bevacizumab doses were ascertained from sites at the time of site initiation. Subjects were treated with all or any components of second-line treatment until the occurrence of unacceptable adverse events, disease progression, death, loss to follow up, or study withdrawal by the subject, investigator, or sponsor. Tumor response was evaluated by blinded central radiology review per modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 and by the investigator using either modified RECIST version 1.0 or clinical assessment. After subjects permanently discontinued all components of second-line treatment, they were to undergo a safety follow-up assessment 30 (± 7) days after the last dose. Subjects ending second-line treatment before disease progression were followed for PFS (radiographic disease assessment) every 12 weeks (± 14 days) from the safety follow-up visit until disease progression, initiation of a new therapy for mCRC, or until approximately 100 PFS events were observed in subjects with wild-type KRAS tumors. Subjects were also followed for survival every 12 weeks (± 14 days) from the safety follow-up assessment until approximately 100 PFS events were observed in subjects with wild-type KRAS tumors.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of metastatic adenocarcinoma of the colon or rectum that cannot, in the opinion of the investigator, be cured by surgical resection at the time of randomization
* Wild-type KRAS expressing mCRC from the primary tumor or metastasis.
* Failure of prior first-line oxaliplatin-based chemotherapy with bevacizumab (at least four therapeutic doses of oxaliplatin-based chemotherapy and bevacizumab) for mCRC.
* At least one uni-dimensionally measurable lesion per modified RECIST criteria.
* Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Man or woman 18 years of age or older
* Hematology, chemistry, coagution, metabolic functions within normal or protocol-defined limits

Exclusion Criteria

* Previous irinotecan, anti-EGFr therapy (eg, cetuximab, panitumumab, erlotinib, gefitinib, lapatinib) or vaccine for the treatment of mCRC
* Radiotherapy ≤ 14 days before randomization
* Evidence of central nervous system (CNS) metastases
* Unresolved toxicities from prior anti-cancer therapy that, in the opinion of the investigator, precludes subject from participation
* History of other invasive primary cancer, except:
* Curatively resected or treated non-melanomatous skin cancer
* Curatively treated cervical carcinoma in situ
* Other primary solid tumor treated curatively and no treatment administered ≤ 2 years before randomization and, in the investigator's opinion, it is unlikely that there will be a recurrence ≤ 2 years post randomization

Medications

* C hronic daily treatment (as determined by the investigator) with aspirin (> 325 mg/day) or non steroidal anti inflammatory agents known to inhibit platelet function
* Infection requiring a course of systemic anti-infectives that was completed ≤ 14 days before randomization (exception can be made at the judgment of the investigator for oral treatment of an uncomplicated urinary tract infection [UTI])
* Subjects concurrently receiving any investigational agent or therapy ≤ 30 days before randomization

General:

* Significant cardiovascular risk as defined by the protocol
* History of peripheral arterial ischemia ≤ 24 weeks before randomization (subjects with brief, reversible, exercise-induced claudication are eligible)
* History of visceral arterial ischemia ≤ 24 weeks before randomization
* Significant bleeding risk:
* Major surgical procedure, open biopsy, or significant traumatic injury ≤ 28 days before randomization
* Anticipation of need for major surgical procedures during the course of the study
* C ore biopsy or other minor procedure, excluding placement of a vascular access device ≤ 7 days before randomization
* A ny significant bleeding that is not related to the primary colon tumor ≤ 24 weeks before randomization
* P re-existing bleeding diathesis or coagulopathy with the exception of well-controlled chronic anticoagulation therapy
* Serious or non-healing wounds, skin ulcers, or unhealed bone fractures
* Gastroduodenal ulcer(s) determined by endoscopy to be active or uncontrolled gastrointestinal ulcer ≤ 28 days before randomization
* History of interstitial lung disease (eg, pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest x-ray (CXR) or computed tomography (CT) scan
* Clinically significant ascites
* Subjects known to be human immunodeficiency virus (HIV) positive or known to have chronic or active hepatitis B or C infection
* Men and women of childbearing potential (women who are post-menopausal < 52 weeks, not surgically sterilized, or not abstinent) who do not consent to use adequate contraception (according to institutional standard of care) during the course of the study and after the last date of receiving second-line treatment (24 weeks for women, 4 weeks for men)
* Women who test positive for serum or urine pregnancy test ≤ 72 hours before randomization or are breast-feeding
* Subjects allergic to any component that is part of the treatment regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2012-05-10 (Actual); Study Completion 2013-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Hecht JR, Cohn A, Dakhil S, Saleh M, Piperdi B, Cline-Burkhardt M, Tian Y, Go WY. SPIRITT: A Randomized, Multicenter, Phase II Study of Panitumumab with FOLFIRI and Bevacizumab with FOLFIRI as Second-Line Treatment in Patients with Unresectable Wild Type KRAS Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2015 Jun;14(2):72-80. doi: 10.1016/j.clcc.2014.12.009. Epub 2015 Jan 8. PMID 25982297
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We enrolled 266 subjects, but we only perform analyses on the Full Analysis Set, defined as all randomized subjects who provide informed consent before the initiation of any study specific procedures and who receive at least one dose of panitumumab or bevacizumab. There are 264 patients in this Full Analysis Set.
Groups:
- Panitumumab Plus FOLFIRI: subjects in this arm receive once-every-2-weeks (Q2W) FOLFIRI regimen plus panitumumab 6 mg/kg
- Bevacizumab Plus FOLFIRI: subjects in this arm receive once-every-2-weeks (Q2W) FOLFIRI regimen plus bevacizumab (either 5 mg/kg or 10 mg/kg, depending on physician choice and institutional standard of care)
Period: Overall Study
Arm/Group | Panitumumab Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Started | 133 | 131
Completed | 109 | 108
Not Completed | 24 | 23
Not completed — Reimbursement | 1 | 0
Not completed — Administrative decision | 3 | 3
Not completed — Withdrawal by Subject | 16 | 15
Not completed — Lost to Follow-up | 1 | 3
Not completed — Adverse Event | 1 | 1
Not completed — On-going | 1 | 1
Not completed — Ineligibility Determined | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panitumumab Plus FOLFIRI | Bevacizumab Plus FOLFIRI | Total
Number analyzed (Participants) | 133 | 131 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.6) | 59.1 (9.9) | 59.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 92
  Male | 87 | 85 | 172
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 102 | 95 | 197
  Black or African American | 21 | 18 | 39
  Hispanic or Latino | 5 | 9 | 14
  Asian | 4 | 8 | 12
  American Indian or Alaska Native | 1 | 0 | 1
  Other | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — Scale range from 0 (fully active) to 5(dead), only status 0 or 1 is included by protocol.
  Participants
    0 (Fully active) | 74 | 70 | 144
    1 (Restricted in physically strenuous activity) | 58 | 61 | 119
    Missing | 1 | 0 | 1
Primary tumor diagnosis [Number; unit: Participants]
  Colon | 102 | 91 | 193
  Rectum | 31 | 40 | 71
Number of metastatic organs [Number; unit: Participants]
  1 | 49 | 61 | 110
  2 | 39 | 42 | 81
  >=3 | 44 | 28 | 72
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as time from the date of randomization to the date of first progression per modified RECIST version 1.0 (based on central review of the radiographic scans), or death within 60 days after the last evaluable tumor assessment or randomization date (whichever is later).
Time Frame: From randomization up to 65 months.
Population: Analysis population include all enrolled subjects who received at least one dose of study therapy and do not include subjects with unevaluable KRAS status.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Number analyzed (Participants) | 127 | 123
months
  Wild-type KRAS (n=91,91) | 7.7 [5.7 to 11.8] | 9.2 [7.8 to 10.6]
  Mutant KRAS (n=36,32) | 3.7 [2.7 to 5.5] | 6.4 [3.5 to 17.1]

2. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from the date of randomization to the date of death due to any cause. Subjects who have not died or are lost to follow-up at the analysis cutoff date will be censored at their last contact date.
Time Frame: From randomization up to 65 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Number analyzed (Participants) | 127 | 123
months
  Wild-type KRAS (n=91,91) | 18.0 [13.5 to 21.7] | 21.4 [16.5 to 24.6]
  Mutant KRAS (n=36,32) | 8.7 [6.1 to 14.5] | 13.5 [9.1 to 14.3]

3. Secondary Outcome: Objective Response Rate
Description: Objective response rate is defined as incidence of either a confirmed complete response (CR) or partial response (PR) on study up to starting a new anti-tumor therapy and will be based on modified RECIST version 1.0 (responder) by central assessment.
Time Frame: From randomization up to 65 months.
Population: Analysis population include all enrolled subjects who received at least one dose of study therapy, who had at least one baseline uni-dimensionally measurable target lesion based on central (and investigator, respectively) assessment using a modified RECIST criteria version 1.0, and who had evaluable KRAS status.
Measure: Number (95% Confidence Interval); unit: % of patients
Arm/Group | Panitumumab Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Number analyzed (Participants) | 121 | 113
% of patients
  Wild-type KRAS (n=91,91) | 32.18 [22.56 to 43.06] | 19.28 [11.44 to 29.41]
  Mutant KRAS (n=36,32) | 11.76 [3.30 to 27.45] | 3.33 [0.08 to 17.22]

4. Secondary Outcome: Time to Response
Description: Time to response is defined as time from the date of randomization to the date of first confirmed objective response
Time Frame: From randomization up to 65 months.
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Panitumumab Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Number analyzed (Participants) | 121 | 113
months
  Wild-type KRAS (n=91,91) | 2.1 (2.2) [1.8 to 3.9] | 3.7 (1.2) [2.0 to 4.0]
  Mutant KRAS (n=36,32) | 2.2 (0.2) [2.0 to 2.3] | 1.8 (NA) [1.8 to 1.8]

5. Secondary Outcome: Time to Progression
Description: Time to progression is defined as time from the date of randomization to the date of radiographic disease progression per modified RECIST version 1.0 (per central assessment).
Time Frame: From randomization up to 65 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Number analyzed (Participants) | 127 | 123
months
  Wild-type KRAS | 11.1 [7.5 to 13.2] | 9.4 [8.2 to 11.9]
  Mutant KRAS | 4.5 [3.0 to 12.0] | 7.4 [5.7 to 19.2]

6. Secondary Outcome: Disease Control
Description: Disease control is defined as incidence of objective response or stable disease on study up to starting a new anti-tumor therapy.
Time Frame: From randomization up to 65 months.
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Panitumumab Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Number analyzed (Participants) | 121 | 113
% of participants
  Wild-type KRAS (n=91,91) | 72.41 [61.79 to 81.46] | 79.52 [69.24 to 87.59]
  Mutant KRAS (n=36,32) | 52.94 [35.13 to 70.22] | 66.67 [47.19 to 82.71]

7. Secondary Outcome: Duration of Response
Description: Duration of response is defined as time from first confirmed objective response to disease progression per modified RECIST version 1.0 (by central assessment).
Time Frame: From randomization up to 65 months.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Number analyzed (Participants) | 121 | 113
months
  Wild-type KRAS (n=91,91) | 12.7 [7.9 to 19.1] | 8.9 [6.5 to 13.6]
  Mutant KRAS (n=36,32) | 10.2 [9.8 to 13.5] | 15.2 [NA to NA] — Only 1 event of response in this category.

ADVERSE EVENTS:
Time Frame: The median reporting period was since randomization date to 65 months.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  Summary of Adverse Events includes only those subjects who received at least one dose of investigational product.
Arm/Group | Panitumumab Plus FOLFIRI | Bevacizumab Plus FOLFIRI
Serious Adverse Events (participants affected / at risk) | 61/133 | 39/131
Other Adverse Events (participants affected / at risk) | 133/133 | 129/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus FOLFIRI (N=133) | Bevacizumab Plus FOLFIRI (N=131)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 4
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal ulcer (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 5 | 3
Vomiting projectile (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 2 | 1
Chest pain (General disorders) | 1 | 1
Device occlusion (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Stent malfunction (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 3 | 2
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 3
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Heart injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 6
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 2 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus FOLFIRI (N=133) | Bevacizumab Plus FOLFIRI (N=131)
Anaemia (Blood and lymphatic system disorders) | 28 | 30
Leukopenia (Blood and lymphatic system disorders) | 11 | 14
Neutropenia (Blood and lymphatic system disorders) | 44 | 53
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 19
Conjunctivitis (Eye disorders) | 11 | 3
Lacrimation increased (Eye disorders) | 10 | 6
Abdominal pain (Gastrointestinal disorders) | 23 | 37
Abdominal pain upper (Gastrointestinal disorders) | 11 | 4
Constipation (Gastrointestinal disorders) | 43 | 34
Diarrhoea (Gastrointestinal disorders) | 93 | 87
Dyspepsia (Gastrointestinal disorders) | 13 | 12
Flatulence (Gastrointestinal disorders) | 7 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 9
Nausea (Gastrointestinal disorders) | 69 | 88
Stomatitis (Gastrointestinal disorders) | 41 | 33
Vomiting (Gastrointestinal disorders) | 47 | 47
Asthenia (General disorders) | 9 | 18
Chills (General disorders) | 9 | 7
Fatigue (General disorders) | 76 | 80
Mucosal inflammation (General disorders) | 35 | 30
Oedema peripheral (General disorders) | 17 | 10
Pain (General disorders) | 10 | 7
Pyrexia (General disorders) | 21 | 13
Paronychia (Infections and infestations) | 14 | 0
Upper respiratory tract infection (Infections and infestations) | 15 | 15
Urinary tract infection (Infections and infestations) | 12 | 15
International normalised ratio increased (Investigations) | 7 | 1
Weight decreased (Investigations) | 26 | 35
Weight increased (Investigations) | 7 | 1
Decreased appetite (Metabolism and nutrition disorders) | 38 | 41
Dehydration (Metabolism and nutrition disorders) | 28 | 25
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 42 | 23
Hypomagnesaemia (Metabolism and nutrition disorders) | 47 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 15
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 12
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 7
Dizziness (Nervous system disorders) | 17 | 12
Dysgeusia (Nervous system disorders) | 6 | 9
Headache (Nervous system disorders) | 11 | 12
Neuropathy peripheral (Nervous system disorders) | 11 | 19
Anxiety (Psychiatric disorders) | 12 | 8
Depression (Psychiatric disorders) | 11 | 9
Insomnia (Psychiatric disorders) | 20 | 21
Proteinuria (Renal and urinary disorders) | 0 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 29
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 28
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 36 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 | 9
Nail disorder (Skin and subcutaneous tissue disorders) | 13 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 7
Rash (Skin and subcutaneous tissue disorders) | 80 | 9
Skin fissures (Skin and subcutaneous tissue disorders) | 16 | 2
Deep vein thrombosis (Vascular disorders) | 8 | 1
Hypertension (Vascular disorders) | 2 | 11
Hypotension (Vascular disorders) | 19 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.